CLINICAL TRIAL: NCT01771458
Title: A Randomized Proof-of-concept Phase II Trial Comparing Therapy Based on Tumor Molecular Profiling Versus Conventional Therapy in Patients With Refractory Cancer.
Brief Title: A Randomized Phase II Trial Comparing Therapy Based on Tumor Molecular Profiling Versus Conventional Therapy in Patients With Refractory Cancer
Acronym: SHIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IC 2012-04
Record Dates: First submitted 2012-11-27; First posted 2013-01-18 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Reccurent/Metastatic Solid Tumor Disease
Keywords: Metastatic/Reccurent; Solid Tumor; Refractory; Molecular profile; Targeted treatment
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard chemotherapy (Active Comparator): Treatment choice is based on Investigator decision.
  Interventions: Procedure: Tumor biopsy; Drug: Standard Chemotherapy
- Personalized treatment (Experimental): Targeted therapy based on the patient molecular profil (if there is at least one abnormality that could be targeted)
  Elligible therapies in this trial are :
  Imatinib Everolimus Vemurafenib Sorafenib Erlotinib Lapatinib Trastuzumab Dasatinib Tamoxifen (or letrozole if contra-indication) Abiraterone
  Interventions: Drug: Targeted therapy based on molecular profiling : Imatinib; Procedure: Tumor biopsy; Drug: Targeted therapy based on molecular profiling : Everolimus; Drug: Targeted therapy based on molecular profiling : Vemurafenib; Drug: Targeted therapy based on molecular profiling : Sorafenib; Drug: Targeted therapy based on molecular profiling : Erlotinib; Drug: Targeted therapy based on molecular profiling : Lapatinib + Trastuzumab; Drug: Targeted therapy based on molecular profiling : Dasatinib; Drug: Targeted therapy based on molecular profiling : Tamoxifen (or letrozole if contra-indication); Drug: Targeted therapy based on molecular profiling : Abiraterone

INTERVENTIONS:
Drug: Targeted therapy based on molecular profiling : Imatinib
  Arms: Personalized treatment
Procedure: Tumor biopsy
Drug: Standard Chemotherapy
  Other Names: Based on each investigator choice
  Arms: Standard chemotherapy
Drug: Targeted therapy based on molecular profiling : Everolimus
  Arms: Personalized treatment
Drug: Targeted therapy based on molecular profiling : Vemurafenib
  Arms: Personalized treatment
Drug: Targeted therapy based on molecular profiling : Sorafenib
  Arms: Personalized treatment
Drug: Targeted therapy based on molecular profiling : Erlotinib
  Arms: Personalized treatment
Drug: Targeted therapy based on molecular profiling : Lapatinib + Trastuzumab
  Arms: Personalized treatment
Drug: Targeted therapy based on molecular profiling : Dasatinib
  Arms: Personalized treatment
Drug: Targeted therapy based on molecular profiling : Tamoxifen (or letrozole if contra-indication)
  Arms: Personalized treatment
Drug: Targeted therapy based on molecular profiling : Abiraterone
  Arms: Personalized treatment

SUMMARY:
SHIVA is a proof of concept randomized phase II trial which compares two treatment strategies for patients with refractory cancer.

From a tumor biopsy, a molecular profile of the disease is established (mutations, amplifications, hormone receptor status). If a molecular abnormality is identified for which an approved targeted agent is available, patients are randomized randomized between two arms:

* Targeted therapy based on the molecular profile
* Conventional therapy based on investigator's choice.

A cross-over is proposed at disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with recurrent/metastatic solid tumor who failed or are not candidate for treatments usually proposed in first intentions and for whom a prospective clinical trial has been indicated in a tumor board
2. ECOG performance status of 0 or 1
3. Biopsiable disease (tumor biopsy mandatory for tumor profiling). The biopsy can be performed when patients are being treated with standard therapy for their recurrent/metastatic cancer if it is not planned to treat them with molecularly targeted agents in the future.
4. Measurable disease
5. Adequate renal function defined by a serum creatinine <1.5xUNL (upper normal limit)
6. Adequate liver function test defined by SGOT & SGPT <3xUNL (5xUNL in case of liver metastases), and bilirubin level <1.5xUNL
7. Adequate bone marrow function defined by platelets >100,000/mm3, hemoglobin >10 g/dL, and neutrophils >1,000/mm3
8. Patients must be affiliated to the French Social Security System
9. Signed informed consent
10. For female of child-bearing potential: a negative pregnancy test <72 hours before starting study treatment is required. If sexually active, female of childbearing potential must use "highly effective" methods of contraception for the study duration and for 3 months following the last treatment
11. For male of reproductive potential: any sexually active male patient must use a condom while on study treatment and for 3 months following the last treatment
12. Agreement to send the CD-ROMs of imaging for central review

Exclusion Criteria:

1. Patients who have only bone and/or brain metastases
2. Patients whose brain metastases have not been controlled for >3 months
3. Patient participating in another clinical trial with an experimental drug
4. Patients who are candidate to receive a molecularly targeted agent that is approved for their disease
5. Anticoagulation with anti-vitamin K (Low Molecular Weight Heparin [LMWH] is allowed)
6. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, including uncontrolled diabetes, cardiac disease, uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infection within one year, chronic liver or renal disease, active gastrointestinal tract ulceration, severely impaired lung function
7. Pregnant and/or breastfeeding women
8. Individually deprived of liberty or placed under the authority of a tutor
9. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
10. Known HIV, HBV, or HCV infection

Eligibility criteria for the randomized part :

1. Identification of tumor molecular abnormalities for which the Therapeutic Decision Committee (TDC) recommends a molecularly targeted therapy available in the context of the trial (even if the molecular profile is incomplete)
2. Therapy recommended by the TDC is not approved for the patient's disease
3. ECOG performance status of 0 or 1
4. Adequate renal function defined by a serum creatinine <1.5xUNL
5. Adequate liver function tests defined by SGOT & SGPT <3xUNL (5xUNL in case of liver metastases), and bilirubin level <1.5xUNL
6. Adequate bone marrow function defined by platelets >100,000/mm3, hemoglobin >8 g/dL, and neutrophils >1,000/mm3
7. Albumin, LDH and number of metastatic sites have been documented (in order to determine the RMH prognostic score)
8. LVEF >50%
9. QTc <480 ms on ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient's progression free survival (according RECIST 1.1) of targeted therapy based on molecular profiling versus conventional chemotherapy.
  Tumor evaluation according to RECIST 1.1 criteria (every 2 months)

SECONDARY OUTCOMES:
Overall response rate (ORR)
  Tumor evaluation according to RECIST 1.1 criteria (every 2 months)
Overall Survival (OS)
Treatments side effects assessement according to the NCI CTCAE v4.03 scale.
Treatment effect variations as defined by tumor growth according to the altered signaling pathway
  Evaluation of tumor growth before and during the study (according to RECIST 1.1)
Patient's progression free survival (according RECIST 1.1) of targeted therapy based on molecular profiling versus conventional chemotherapy after cross-over.
  Tumor evaluation according to RECIST 1.1 criteria (every 2 months)
Evaluation of the ability of ctDNA to early predict treament efficacy
  Comparing treatment efficacy to ctDNA level (before and during treatment course)
Evaluation of the medico-economic impact of the experimental strategy
Technical feasability of the SHIVA trial: number of screened patient compared to number of patients elligible to randomization.
  Number of screened patients. Number of patient with a molecular full profil in the timeframe (4 weeks between tumor biopsy and SHIVA's committees decision).
  Number of randomized patient.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LE TOURNEAU, MD, Principal Investigator — Institut Curie
Locations (8):
- France (8):
  - Centre régional de lutte contre le cancer de Bourgogne Georges François Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Insitut Curie, Paris
  - Institut Curie Hopital Rene Huguenin, Saint-Cloud
  - Institut de cancérologie de l'Ouest Centre René Gauducheau, Saint-Herblain
  - Institut Claudius Régaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Belin L, Kamal M, Mauborgne C, Plancher C, Mulot F, Delord JP, Goncalves A, Gavoille C, Dubot C, Isambert N, Campone M, Tredan O, Ricci F, Alt M, Loirat D, Sablin MP, Paoletti X, Servois V, Le Tourneau C. Randomized phase II trial comparing molecularly targeted therapy based on tumor molecular profiling versus conventional therapy in patients with refractory cancer: cross-over analysis from the SHIVA trial. Ann Oncol. 2017 Mar 1;28(3):590-596. doi: 10.1093/annonc/mdw666. PMID 27993804
- [Derived] Le Tourneau C, Delord JP, Goncalves A, Gavoille C, Dubot C, Isambert N, Campone M, Tredan O, Massiani MA, Mauborgne C, Armanet S, Servant N, Bieche I, Bernard V, Gentien D, Jezequel P, Attignon V, Boyault S, Vincent-Salomon A, Servois V, Sablin MP, Kamal M, Paoletti X; SHIVA investigators. Molecularly targeted therapy based on tumour molecular profiling versus conventional therapy for advanced cancer (SHIVA): a multicentre, open-label, proof-of-concept, randomised, controlled phase 2 trial. Lancet Oncol. 2015 Oct;16(13):1324-34. doi: 10.1016/S1470-2045(15)00188-6. Epub 2015 Sep 3. PMID 26342236